Investigating the Effectiveness of an Entertainment Education Short Film for Internalized HIV Stigma Reduction, Intimate Partner Status Disclosure Intentions, and Antiretroviral Medical Adherence Intentions: A Randomized Controlled Trial Among Black Women Living with HIV in the Southern U.S.

ClinicalTrials.Gov Identifier: NCT03898063

April 1, 2020

Study #: 20170967 Effective Date: 4/1/2020

# **University of Miami**

# CONSENT TO PARTICIPATE IN A RESEARCH STUDY 90 Days Study

The following information describes the research study in which you are being asked to take part. Please read this carefully. At the end, you will be asked if you agree.

## **PURPOSE OF STUDY**

You are being asked to be in a research study. The purpose of this study is to get your thoughts about the short film, *90 Days*. We also want to know about your thoughts about HIV/AIDS stigma, medical adherence and chats about HIV/AIDS with sexual partners.

#### **PROCEDURES**

Once you are screened for eligibility, you will fill out two questionnaires. The first survey will ask questions about you, HIV/AIDS, stigma, medical adherence, and disclosure. After completing survey one, you will either read a brochure or watch the short film, 90 Days. Next, you will complete another brief survey about the film or brochure, you, HIV/AIDS, stigma, medical adherence, and disclosure. Altogether, this will take about 35-45 minutes of your time. This study must be completed in one setting.

## **RISKS AND/OR DISCOMFORTS**

We do not expect you will have any discomfort from being in this study. However, it is possible that you may experience some stress in completing the questionnaires. If at any time you feel uncomfortable, you can skip any of the survey questions. You can also end your participation at any time without penalty.

#### **BENEFITS**

No direct benefit can be promised to you from being in this study.

#### CONFIDENTIALITY

The pre- and post-film surveys will not ask any information that can identify you.

# **COMPENSATION**

After completing the pre-survey, the intervention and post-survey, you will be compensated in the amount agreed upon by your panel provider.

## RIGHT TO DECLINE OR WITHDRAW

Being in this study is voluntary. You are free to say no or leave at any time during the study.

## **CONTACT INFORMATION**

The direct contact for this study is Jazmyne Simmons (<u>jvs11@miami.edu</u>). Also, the principal investigator, Dr. Nick Carcioppolo (305-284-5633) will gladly answer any questions you may have about the this project. If you have questions about your rights

- Study #: 20170967 Effective Date: 4/1/2020

# **University of Miami**

# CONSENT TO PARTICIPATE IN A RESEARCH STUDY 90 Days Study

as a research participant, you may contact the Human Subjects Research Office at the University of Miami at (305) 243-3195.

# **PARTICIPANT AGREEMENT**

I have read the information in this consent form and agree to participate. Clicking "Yes, I consent to participate" below will be considered your informed consent to participate and record your anonymous responses in this research study: